CLINICAL TRIAL: NCT00188877
Title: A Phase II Study of Intensity Modulated Radiation Therapy for Nasopharyngeal Cancer
Brief Title: Intensity Modulated Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 03-0158-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Procedure: intensity modulated radiation therapy
Drug: cisplatinium and fluorouracil - standard treatment

SUMMARY:
Many normal tissues, including the eyes, brain, and spinal cord are very close to cancers in the nasopharynx. The dose of radiation delivered to the cancer is limited by tolerance of these normal tissues. Standard radiation treatment techniques using three or four radiation beams cannot avoid delivering some dose of radiation to these normal tissues that do not need to get radiation. Intensity Modulated Radiation Therapy (IMRT) uses many hundreds of computer-controlled radiation beams aimed at your cancer to try to lower the amount of radiation that normal tissues receive, while still delivering the desired amount of radiation to your cancer and to areas that your doctor thinks may have cancer cells.

The doctors at Princess Margaret Hospital are conducting this study in order to test whether the use of IMRT techniques can improve the chance of controlling your cancer in the head and neck region.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histopathologic diagnosis of nasopharyngeal squamous cell carcinoma requiring primary radiation
* less than 70 yrs of age
* Stage T1-T4; N0-N3; M0
* KPS less than 70
* no prior RT to H&N or chemotherapy for H&N
* no other malignancy except non-melanomatous skin cancer
* no distant mets
* no contraindication to RT or chemotherapy
* adequate organ function
* informed consent

Exclusion Criteria

* Major medical or psychiatric illness, which would interfere with either completion of therapy and follow-up or with full and complete understanding of the risks and potential complications of the therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2003-06 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate 3 year local progression free survival in patients with nasopharyngeal carcinoma treated with Intensity Modulated Radiation Therapy (IMRT) techniques. | q2 monthly during year 1, q3 monthly during year 2; q4 monthly during year 3; q6 monthly during year 4 and annually thereafter

SECONDARY OUTCOMES:
-the ability of IMRT techniques to spare long term xerostomia as evaluated by saliva flow rates.
-the nature and prevalence of acute and late side effects and their relationship to local dose.
-the dosimetric differences between conventional "forward planned" two dimensional plans, three dimensional plans and Intensity modulated radiation therapy.
-evaluation of failure with respect to the doses in the region of the failure
-quality of life measurements in patients after receiving IMRT for the treatment of nasopharyngeal carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bayley, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada